CLINICAL TRIAL: NCT01521494
Title: PA21 Phase II Clinical Study in Hemodialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA1201
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- PA21 750 mg/day (Experimental)
  Interventions: Drug: PA21
- PA21 1500 mg/day (Experimental)
  Interventions: Drug: PA21
- PA21 2250 mg/day (Experimental)
  Interventions: Drug: PA21
- PA21 3000 mg/day (Experimental)
  Interventions: Drug: PA21
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PA21
  Arms: PA21 750 mg/day
Drug: PA21
  Arms: PA21 1500 mg/day
Drug: PA21
  Arms: PA21 2250 mg/day
Drug: PA21
  Arms: PA21 3000 mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate dose-response efficacy and safety in hemodialysis patients with hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 20 or older, regardless of gender.
* Receiving stable maintenance hemodialysis 3 times a week.
* Patients not having changed their phosphate binder agent dose, for 4 weeks or more before their observation period start.

Exclusion Criteria:

* Patients having history of a pronounced brain / cardiovascular disorder.
* Patients having severe gastrointestinal disorders.
* Patients having severe hepatic disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2012-07-03 (Actual); Study Completion 2012-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Clinical Development Department, Kissei pharmaceutical Co., Ltd.
Locations (1):
- Japan, Multiple Locations, Japan

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21 750 mg/Day; PA21 1500 mg/Day; PA21 2250 mg/Day; PA21 3000 mg/Day: PA21
- Placebo: Placebo
Period: Overall Study
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo
Started | 39 | 36 | 35 | 36 | 37
Completed | 37 | 31 | 23 | 15 | 30
Not Completed | 2 | 5 | 12 | 21 | 7
Not completed — Adverse Event | 1 | 2 | 9 | 6 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 0
Not completed — Decrease in serum phosphate | 0 | 2 | 3 | 12 | 0
Not completed — Decrease in serum calcium | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Total of 5 patients were excluded from analysis because they failed to have primary endpoint.
Groups:
- Total: Total of all reporting groups
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo | Total
Number analyzed (Participants) | 39 | 35 | 33 | 34 | 37 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (10.4) | 63.8 (12.0) | 61.9 (10.5) | 61.4 (11.2) | 60.8 (10.2) | 61.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 15 | 14 | 63
  Male | 27 | 23 | 23 | 19 | 23 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 39 | 35 | 33 | 34 | 37 | 178
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Dialysis vintage [Mean (Standard Deviation); unit: months] | 77.6 (67.5) | 85.1 (60.7) | 95.8 (81.9) | 91.5 (58.6) | 71.0 (45.0) | 83.7 (63.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Phosphorus Concentrations at the End of Treatment.
Description: Changes in serum phosphorus concentrations from baseline to the end of treatment were adjusted by serum phosphorus concentration at baseline.
Time Frame: 6 weeks
Population: Total of 5 patients were excluded from analysis because they failed to have primary endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo
Number analyzed (Participants) | 39 | 35 | 33 | 34 | 37
mg/dL | -1.84 [-2.23 to -1.44] | -2.59 [-3.01 to -2.17] | -3.17 [-3.60 to -2.74] | -3.78 [-4.20 to -3.36] | 0.14 [-0.26 to 0.55]

2. Secondary Outcome: Change From Baseline in Serum Calcium Concentrations.
Time Frame: 6 weeks
Population: Total of 5 patients were excluded from analysis because they failed to have primary endpoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo
Number analyzed (Participants) | 39 | 35 | 33 | 34 | 37
mg/dL | 0.20 (0.34) | 0.16 (0.33) | 0.38 (0.44) | 0.38 (0.39) | -0.09 (0.31)

3. Secondary Outcome: Change From Baseline in Serum Intact-PTH Concentrations.
Time Frame: 6 weeks
Population: Some patients were excluded from analysis because they failed to have primary endpoint or missed to measure intact-PTH at the end of treatment.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo
Number analyzed (Participants) | 39 | 34 | 31 | 31 | 37
pg/mL | -35.2 (89.8) | -45.6 (79.2) | -97.0 (92.7) | -86.5 (104.0) | 21.5 (82.5)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | PA21 750 mg/Day | PA21 1500 mg/Day | PA21 2250 mg/Day | PA21 3000 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36 | 0/35 | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/39 | 2/36 | 2/35 | 1/36 | 1/37
Other Adverse Events (participants affected / at risk) | 13/39 | 11/36 | 19/35 | 20/36 | 11/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 750 mg/Day (N=39) | PA21 1500 mg/Day (N=36) | PA21 2250 mg/Day (N=35) | PA21 3000 mg/Day (N=36) | Placebo (N=37)
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 750 mg/Day (N=39) | PA21 1500 mg/Day (N=36) | PA21 2250 mg/Day (N=35) | PA21 3000 mg/Day (N=36) | Placebo (N=37)
Nasopharyngitis (Infections and infestations) | 5 | 5 | 3 | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 13 | 15 | 7
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No